CLINICAL TRIAL: NCT01379807
Title: A Phase II Trial to Assess the Efficacy and Safety of Panitumumab Combined With Docetaxel and Cisplatin as a First-line Treatment of Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Efficacy and Safety of Panitumumab Combined With Docetaxel and Cisplatin as a First-line Treatment of Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Acronym: SPIGA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Gallego de Investigaciones Oncologicas (Other)
Collaborators: Amgen (Industry); Trial Form Support S.L. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GGIO-2010-01
Record Dates: First submitted 2011-06-22; First posted 2011-06-23 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2011-04

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Panitumumab; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- panitumumab + docetaxel + cisplatino (Experimental)
  Interventions: Drug: panitumumab + docetaxel + cisplatino

INTERVENTIONS:
Drug: panitumumab + docetaxel + cisplatino — Panitumumab, docetaxel and cisplatin combination treatment will be administered for 6 months or until disease progression (PD) according to investigator's criteria unacceptable toxicity or consent withdrawal.

SUMMARY:
The clinical hypothesis of this study is that the addition of Panitumumab to the first line treatment combination of docetaxel plus cisplatin will provide benefit to patients with advanced gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent Inclusion:
* Age ≥ 18 years
* Histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction with advanced unresectable or metastatic disease.
* Measurable disease per the revised RECIST (Response Evaluation Criteria in Solid Tumor) Guidelines
* ECOG performance score of 0 - 2
* Within seven days prior to initiating study treatment:Haematology:Neutrophils ≥ 1.5x109, Platelets ≥ 100x10/ L, Hemoglobin ≥ 9g/dL. Hepatic functions: Total bilirubin ≤ 1.5 time the upper normal limit (UNL),ASAT ≤ 2.5xUNL in absence of liver metastases, or ≤5xUNL in presence of liver metastases,ALAT ≤ 2.5xUNL in absence of liver metastases, or ≤5xUNL in presence of liver metastases. Renal function: creatinine clearance ≥50 mL/min. Metabolic Function: Magnesium ≥ lower limit of normal, Calcium ≥ lower limit of normal.

Exclusion Criteria:

* Prior chemotherapy or other anticancer therapy for advanced unresectable or metastatic disease (1st line)
* Prior anti-EGFR antibody therapy (e.g. cetuximab) or treatment with small molecule EGFR inhibitors (e.g. erlotinib).
* HER2-positive tumor (centrally assessed)
* Past or current history (within the last 5 years prior to treatment start) of other malignancies except gastric cancer (Patients with curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible)
* Current or prior history of central nervous system metastases
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications Treatment with any other investigational agent, or participation in another clinical trial within 30 days prior to entering this study
* Known hypersensitivity to any of the study drugs
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrollment
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 years
  To estimate the objective response rate in patients treated with docetaxel, cisplatin and panitumumab as first-line treatment in advanced gastric or gastroesophageal junction adenocarcinoma.

SECONDARY OUTCOMES:
Disease control rate | 3 years
Duration of response | 3 years
Time to response | 3 years
Time to progression | 3 years
Time to treatment failure | 3 years
Duration of stable disease | 3 years
Progression free survival | 3 years
Overall survival | 3 years
Safety profile | 3 years
  To describe the safety profile of this combination therapy in the 1st-line setting including the incidence of AE's and changes in laboratory parameters.
Exploratory Objectives | 3 years
  To investigate the predictive potential of different biomarkers on efficacy and/or safety endpoints.

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Complejo Hospitalario Universitario de A Coruña, A Coruña, La Coruña
  - Centro Oncológico de Galícia, A Coruña, La Coruña
  - Hospital Arquitecto Mercide, Ferrol, La Coruña
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, La Coruña
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Complejo Hospitalario Ourense, Ourense, Ourense
  - Hospital de Pontevedra, Pontevedra, Pontevedra
  - Complejo Hospitalario Universitario de Vigo (Xeral Cies), Vigo, Pontevedra
  - Policlínica de Vigo S.A., Vigo, Pontevedra